CLINICAL TRIAL: NCT04117867
Title: The Association Between Intraoperative Hypotension and Perioperative Stroke in General Surgery Patients: a Retrospective, Hospital-based Study in China
Brief Title: The Association Between Intraoperative Hypotension and Perioperative Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Other Study IDs: IOHPS
Record Dates: First submitted 2019-09-27; First posted 2019-10-07 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Perioperative Complication; Intraoperative Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intraoperative hypotension
  Interventions: Behavioral: Patiens with intraoperative hypotension

INTERVENTIONS:
Behavioral: Patiens with intraoperative hypotension — In this study, we will use four previously defined thresholds for intraoperative hypotension: two absolute thresholds (MAP less than 50 mmHg and MAP less than 60 mmHg) and two relative thresholds to the baseline MAP (a decrease of 30% or more and a decrease of 40% or more). A definition of baseline value most frequently reported was the arterial blood pressure before the induction of anesthesia. Therefore, the baseline MAP used in calculating the relative thresholds is defined as the mean MAP of all available blood pressure measurements before induction of anesthesia in the operating room.

SUMMARY:
The aim of this study is to investigate the association between the severity and duration of intraoperative hypotension and the incidence of perioperative stroke after non-cardiac and non-neurologic surgeries.The secondary aim of this study is to confirm the potential risk factors of the perioperative stroke.

DETAILED DESCRIPTION:
Optimized intraoperative management may play an important role in perioperative stroke prevention. Maintaining blood pressure near preoperative baseline values may help decrease the incidence of stroke, however the related evidence is limited.Therefore, this study is to investigate the association between intraoperative hemodynamic variable and the risk of perioperative stroke after non-cardiac and non-neurologic surgeries. The secondary aim of this study is to establish the potential risk factors of the perioperative stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwent surgeries in First hospital affiliated to Shandong First Medical University from January 2013 to October 2019
2. Age>18 or older

Exclusion Criteria:

1. Patients received local infiltration anesthesia
2. Patients underwent total intravenous anesthsia without tracheal intubation or Laryngeal Mask Airway insertion
3. Major vascular operation
4. Neurologic surgery
5. Cariac surgery
6. Intraoperative blood pressure measurements or postoperative neuroimagings measurements are not available
7. History of severe neurological or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent surgical procedures under anesthesia at Qianfoshan Hospital, First Hospital affiliated to Shandong First Medical University during the period from January, 2013, to October, 2019, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative stroke | Within 24 hours after surgery
  Perioperative stroke diagnosed with CT or MRI examination, symptoms and signs
Incidence of perioperative stroke | Within 3 days after surgery
  Perioperative stroke diagnosed with CT or MRI examination, symptoms and signs
Incidence of perioperative stroke | Within 7 days after surgery
  Perioperative stroke diagnosed with CT or MRI examination, symptoms and signs
Incidence of perioperative stroke | Within 30 days after surgery
  Perioperative stroke diagnosed with CT or MRI examination, symptoms and signs

SECONDARY OUTCOMES:
Rate of death | Within 24 hours after surgery
  Death from any cause
Rate of death | Within 3 days after surgery
  Death from any cause
Rate of death | Within 7 days after surgery
  Death from any cause
Rate of death | Within 30 days after surgery
  Death from any cause
Expense of Healthe care and social service | Through study completion, an average of 14 days
  The expense of Healthe care and social service that the patients spent in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Yuelan Wang, Doctor, Principal Investigator — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University
Locations (1):
- The First affiliated hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol